CLINICAL TRIAL: NCT06632067
Title: Comparison of Sugammadex and Neostigmine for Time to Extubation in Adult Patients Undergoing Routine Ophthalmic Surgery Under General Anesthesia
Brief Title: Sugammadex and Time to Extubation in Ophthalmic Surgery
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH112-REC3-124
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: General Anesthesia Using Endotracheal Intubation; Ophthalmologic Surgical Procedure; Sugammadex; Neostigmine; Extubation Readiness
Keywords: sugammadex; general anesthesia; ophthalmologic surgical procedures
MeSH Terms: interventions — Sugammadex; Neostigmine; Atropine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- sugammadex: those who use sugammadex for reversal of neuromuscular blockade
  Interventions: Drug: sugammadex
- neostigmine: those who use neostigmine/atroping for reversal of neuromuscular blockade
  Interventions: Drug: Neostigmine + Atropine

INTERVENTIONS:
Drug: sugammadex — sugammadex used for neuromuscular reversal
  Groups: sugammadex
Drug: Neostigmine + Atropine — Neostigmine and Atropine used for neuromuscular reversal
  Groups: neostigmine

SUMMARY:
This study is to invastigate if patients treated with sugammadex compared to neostigmine/atropine would be extubate faster upon emergence of anesthesia.

DETAILED DESCRIPTION:
This is a retrospective case-control study including patients aged 18 years or older who underwent ophthalmic surgeries under general anesthesia with tracheal intubation between 2020 and 2022. Patients who received rocuronium as the sole neuromuscular blocking agent and were maintained with sevoflurane or desflurane and intravenous fentanyl were included. Based on the choice of reversal agent for neuromuscular blockade, patients were divided into two groups: the sugammadex group or the neostigmine group. Patients who underwent emergency surgery or combined surgeries with other specialties were excluded. Patient characteristics, including age, gender, ASA classification, weight, and height, were collected. Anesthesia-related medications were recorded. The time points of anesthesia induction, start and end of surgery, reversal agent administration, and tracheal extubation were documented.

ELIGIBILITY:
Inclusion Criteria:

aged 18 years or older ophthalmic surgeries under general anesthesia with tracheal intubation between 2020 and 2022 received rocuronium as the sole neuromuscular blocking agent maintained with sevoflurane or desflurane and intravenous fentanyl

Exclusion Criteria:

emergency surgery combined surgeries with other specialties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included patients aged 18 years or older who underwent ophthalmic surgeries under general anesthesia with tracheal intubation between 2020 and 2022. Patients who received rocuronium as the sole neuromuscular blocking agent and were maintained with sevoflurane or desflurane and intravenous fentanyl were included. Based on the choice of reversal agent for neuromuscular blockade, patients were divided into two groups: the sugammadex group or the neostigmine group. Patients who underwent emergency surgery or combined surgeries with other specialties were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Time From reversal to extubation | Time From reversal to extubation
  Time From reversal to extubation
Time From the end of surgery to reversal | Time From the end of surgery to reversal
  Time From the end of surgery to reversal

SECONDARY OUTCOMES:
Time From induction to the end of surgery | Time From induction to the end of surgery
  Time From induction to the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ying Chiang, MD, Principal Investigator — China Medical Univerity Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No